CLINICAL TRIAL: NCT05901610
Title: Decision Making in Chronic Pain and Alcohol Use Disorder
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: personnel availability and challenges with eligibility
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Stephen LaConte, Professor, Virginia Polytechnic Institute and State University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VT IRB# 23-561
Record Dates: First submitted 2023-06-02; First posted 2023-06-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Alcohol Use Disorder; Chronic Pain
MeSH Terms: conditions — Alcoholism; Chronic Pain

STUDY DESIGN:
Intervention Model Description: Each participant will receive all interventions throughout the study. Their pain response will be compared after episodic future thinking (EFT) with the control, episodic recent thinking (ERT) and low-intensity focused ultrasound (LIFU) with the control, Sham LIFU.
Who Masked: Participant
Masking Description: Participants will not be informed whether they are receiving the control behavioral intervention and Sham LIFU.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- EFT and LIFU (Other): Participants will generate positive future events they are looking forward to at several time points in the future (e.g., 2 weeks, 1 month, 3 months, 1 year, and 5 years). During the LIFU condition, participants will have an ultrasound transducer placed on their head, where brief ultrasound pulses are delivered to the desired brain area using the imaging collected during visit 1. A small amount of ultrasound gel will be placed on the face of the single-element focused ultrasound transducer. The transducer will then be fitted on the scalp over the desired brain area and held in place with a mechanical arm. Brief pulses (0.2 to 2 seconds; duty cycle 10 - 70%; pulse repetition frequency 100 - 1000 Hz) of low-intensity (< 50 W/cm2 Isppa), sub-thermal ultrasound (0.3 - 0.5 MHz) will be delivered in order to determine the area of activation, as well as the patterns of brain activity generated.
  Interventions: Behavioral: Episodic Future Thinking; Device: Low-intensity Focused Ultrasound
- EFT and Sham LIFU (Other): Participants will generate positive recent past events that have happened to them at several time points in the previous day (e.g., 7pm-10pm, 4pm-7pm, 1pm-4pm, 10am-1pm, and 7am-10am). During Sham LIFU, the device will be set up identically as in real LIFU. However, the device will be turned off.
  Interventions: Behavioral: Episodic Future Thinking; Device: Sham Low-intensity Focused Ultrasound
- CET ad LIFU (Other): Participants will generate positive recent past events that have happened to them at several time points in the previous day (e.g., 7pm-10pm, 4pm-7pm, 1pm-4pm, 10am-1pm, and 7am-10am). During the LIFU condition, participants will have an ultrasound transducer placed on their head, where brief ultrasound pulses are delivered to the desired brain area using the imaging collected during visit 1.
  Interventions: Behavioral: Control Episodic Thinking; Device: Low-intensity Focused Ultrasound

INTERVENTIONS:
Behavioral: Episodic Future Thinking — Participants will generate descriptions of vivid positive future events.
  Other Names: EFT
  Arms: EFT and LIFU; EFT and Sham LIFU
Behavioral: Control Episodic Thinking — Participants will generate descriptions of vivid positive past events.
  Arms: CET ad LIFU
Device: Low-intensity Focused Ultrasound — A transducer device will use focused ultrasound energy to neuromodulate the insular cortex. The participant's brain will be mapped based on information from the CT and MRI scans, and the transducer will deliver brief ultrasound pulses to the insular cortex.
  Other Names: LIFU
  Arms: CET ad LIFU; EFT and LIFU
Device: Sham Low-intensity Focused Ultrasound — All of the same actions done during LIFU will be performed, but the device will be inactive.
  Other Names: Sham LIFU
  Arms: EFT and Sham LIFU

SUMMARY:
The objective of this within-subject study is to test the effects of Episodic Future Thinking (EFT) and Low-intensity Focused Ultrasound (LIFU) interventions on the pain of subjects who have chronic pain and alcohol use disorder(s).

DETAILED DESCRIPTION:
This study will have a within-subject design. Participants will complete a baseline session (S1) and three intervention sessions. Specifically, participants will complete one intervention session consisting of episodic future thinking (EFT) and low-intensity focused ultrasound (LIFU), a second intervention session consisting of EFT and a control condition for LIFU ("sham-LIFU"), and an intervention session consisting of a control condition for EFT, called control episodic thinking (CET) and LIFU. Measures of chronic pain, alcohol valuation, alcohol craving, and delay discounting will be collected before and after each intervention session. The EFT intervention has participants generate positive events and related cues through a researcher-administered interview-based questionnaire. Participants will be asked to think about and describe positive events that could occur at each of the 6 delays in the future (i.e., 1 week, 1 month, 3 months, 1 year, 5 years, and 25 years). During the LIFU condition, participants will have an ultrasound transducer placed on their head, where brief ultrasound pulses are delivered to the desired brain area. CET requires participants to think about and describe positive events that occurred at each of 6 delays in the past (e.g., last night, yesterday in the afternoon, yesterday in the evening, yesterday in the morning, yesterday in the night, and the night before). After generating these cues participants will be asked to read and consider their cues as they complete the measures again that were collected prior to the cue generation. The sham LIFU condition may be active with ultrasound blocking, or inactive so that it would not deliver stimulation. All participants will complete all three intervention sessions. The first day will be the consent, MRI, and CT scans required for the LIFU intervention. The remaining three intervention sessions will occur in a counterbalanced order. The first and second sessions will be separated by 2-3 weeks, and the remaining sessions will be separated by approximately 1 week.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years old or older
2. Report chronic pain
3. Have sufficiently stable self-reported mental and physical health in order to complete the survey
4. Meet DSM-V clinical criteria for alcohol use disorder (i.e., four or more criteria)
5. Not have unmanaged medical or psychiatric conditions the survey

Exclusion Criteria:

1. Claustrophobia (scanning environment may be uncomfortable)
2. Contraindications to MRI: including pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
3. Contraindications to CT: pregnancy
4. Active medical disorder or treatment with potential CNS effects (e.g. Alzheimer's)
5. History of neurologic disorder (e.g. Parkinson's, Epilepsy, or Essential Tremor)
6. History of head injury resulting in loss of consciousness for >10 minutes
7. Failure to provide a Social Security Number or Tax ID number. This is required for tax purposes.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-06-28 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in Delayed Discounting | Before and after each intervention on two days separated by one week (eight times total).
  Delay discounting tasks provide a measure of the temporal window and examine the devaluation of awards as a function of the delay to the receipt. These computerized assessments provide participants with hypothetical choices between smaller amounts of a reward available immediately and a larger amount of a reward after a range of delays (1 day-25 years). Discounting rates will be measured using adjusting amount delay discounting and minute delay discounting tasks. Change in discounting rates will be compared after different interventions are applied.
Changes in Acute Pain Perception | Before and after each intervention on two days separated by one week (eight times total).
  Sensitivity to acute pain will be measured using a thermal stimulus gradually reaching 50 degrees Celsius. Participants will be asked to rate the induced pain on a visual analogue scale ranging from 0 to 10, such that greater score indicates greater pain perception. The ratings from before and after each intervention will be compared.
Changes in Chronic Pain Severity | Before and after each intervention on two days separated by one week (eight times total).
  Pain severity will be measured using a question from the Brief Pain Inventory. This asking requires participants to rate their pain in the last 24h from 0 to 10. Greater scores indicate greater pain severity.

SECONDARY OUTCOMES:
Change in Alcohol Valuation | Before and after each intervention on two days separated by one week (eight times total).
  Intensity and elasticity of alcohol demand will be determined from an alcohol demand curve via an Alcohol Purchase Task. Change in alcohol demand will be compared within-subjects across sessions and between groups.
Change in Alcohol Craving | Before and after each intervention on two days separated by one week (eight times total).
  Participants will be asked to complete an alcohol urges questionnaire. This questionnaire has 8 questions. Each question has a score that ranges from 1 to 7. Questions 2 and 3 have their scores reversed. The overall score ranges from 8 to 56. Greater scores indicate greater craving.

CONTACTS AND LOCATIONS:
Overall Officials: Wynn Legon, PhD, Principal Investigator — Virginia Polytechnic and State University
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States